CLINICAL TRIAL: NCT03645733
Title: Evaluation of the Effect of Cooled Haemodialysis on Cognitive Function in Patients Suffering With End-stage Kidney Disease: Feasibility Study
Brief Title: Evaluation of the Effect of Cooled Haemodialysis on Cognitive Function in Patients Suffering With End-stage KD
Acronym: E-CHECKED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heart of England NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017054MH
Record Dates: First submitted 2018-08-07; First posted 2018-08-24 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Cognitive Impairment
Keywords: Haemodialysis; Kidney Disease; Mental Health; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Kidney Diseases; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The control group will be at the standard dialysate temperature of 36.5 °C (which is the standard of care in the sites), 3 times a week for 12 months. In the intervention group, patients will receive haemodialysis with a dialysate temperature of 35 degree centigrade. The intervention group will start off using a dialysate temperature that is 36 °C. Thereafter the dialysate temperature will be reduced every two week by 0.5 °C until 35 °C or the lowest tolerated temperature reached. Patients who would fail to tolerate the temperature of 35 °C, the lowest tolerated temperature will be carried over to the end of the study. The intervention group is split into 3 brackets, stratified by age group (patients under 55 years of age, 55-75 and above 75). A third group will also be recruited, but not randomised, consisting of the primary carers (family, friends, etc) of the patients in the other two group to measure the burden they feel in caring for a patient with renal problems.
Who Masked: Outcomes Assessor
Masking Description: One nurse, that gives the patients their cognitive questionnaire battery, is masked from knowing which dialysis fluid temperature the patient is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will be at the standard dialysate temperature of 36.5 °C (which is the standard of care in the sites), 3 times a week for 12 months
- Lower Temperature Group (Experimental): These patients will receive haemodialysis with a dialysate temperature of 35 degree centigrade. The intervention group will start off using a dialysate temperature that is 36 °C. Thereafter the dialysate temperature will be reduced every two week by 0.5 °C until 35 °C or the lowest tolerated temperature reached. Patients who would fail to tolerate the temperature of 35 °C, the lowest tolerated temperature will be carried over to the end of the study.
  Interventions: Procedure: Lower Temperature Group
- Caregivers (No Intervention): Patients, who consent for the study, will be asked to identify the most suitable carer to participate in the study who could be approach in person, over the phone or by post as deemed suitable by the research team and convenient by the carer. Patient's permission to contact their identified carer will be recorded. Carers of consenting patients will be approached in the same manner as above after obtaining patients consent to contact their carers. Patients will still be able to take part in the study even if their carer declines consent.

INTERVENTIONS:
Procedure: Lower Temperature Group — Dialysate temperature of 35 degree centigrade. The intervention group will start off using a dialysate temperature that is 36 °C. Thereafter the dialysate temperature will be reduced every two week by 0.5 °C until 35 °C or the lowest tolerated temperature reached.
  Arms: Lower Temperature Group

SUMMARY:
The Investigators aim to perform a feasibility study that will inform the development of a definitive, fully powered, randomised, controlled clinical trial in the future. The main hypothesis that would be tested in this future trial is that patients treated with regular conventional haemodialysis will have a lesser decline in cognitive function and a better quality of life over one year by using cooler dialysis fluid at 35°C, versus a standard dialysis fluid temperature of 36.5°C. This also should reflect in improvements in their abilities for activities of daily living and therefore, reduce carers' burden. If successful the treatment could be universally applied at no extra cost.

DETAILED DESCRIPTION:
Patients with End-Stage Kidney Disease (ESKD) need haemodialysis to remove excess toxins and fluid from the body and maintain life. They also must restrict their fluid intake, take a median of 19 medications and follow a special diet1. In the UK, 26 000 patients receive haemodialysis at a hospital three times a week for around 4 hours at a yearly cost of £636 million. The numbers needing haemodialysis are rising by 7% per year due to an increase in ageing, diabetes, obesity and hypertension. The best form of treatment for kidney failure is kidney transplantation, but there is a shortage of organ donors with older people being least likely to receive a kidney transplant. The average age of dialysis patients in the UK is 65 with 4-year survival expectancy less than 40% - which is worse than for most cancers. The three most common causes of death are cardiovascular disease, infections and cancer with the greatest mortality in the first three months of starting dialysis. Haemodialysis is a huge burden for patients and their family or carers. Most endure unpleasant dialysis-related symptoms and reduced quality-of-life with high rates of depression, cognitive impairment, hospital admissions and social isolation. Unsurprisingly, dialysis patients value quality-of-life more than life expectancy. Several medications currently used at considerable cost to improve survival and quality-of-life have shown no benefit.

High rates of cognitive impairment in dialysis patients are poorly understood Increasing severity of Chronic Kidney Disease (CKD) is associated with a graded increase in prevalence of cognitive impairment and decrease in brain perfusion independent of vascular risk factors. Diagnostic methods vary but recent reviews summarise at least moderate cognitive impairment in 30-70% of dialysis patients. Cognitive impairment in haemodialysis patients is independently associated with higher rates of depression and mortality. To date, no interventions are proven to slow cognitive decline and this poorly understood association was recently reviewed. Co-segregation of atherosclerotic risk factors, cannot entirely account for excess risk. There are multiple factors CKD and haemodialysis specific factors including oxidative stress, malnutrition and inflammation. Haemodialysis allows accumulation of several neurotoxins that reduce brain perfusion and blood-brain barrier integrity.

Intradialytic hypotension is implicated in excessive cognitive impairment Haemodialysis involves cycles of removing varying volumes of fluid, electrolytes and toxins that accumulate between treatments. Hypotension partially results from fluid removal rates exceeding plasma refill rates. Ubiquitous left ventricular hypertrophy and aortic stiffness further lower the threshold for haemodialysis to inflict recurrent multi-organ ischemia-reperfusion injury. Haemodialysis might cause worsening of cognitive impairment by inducing haemodynamic instability, fluid shifts, cerebral ischaemia or cerebral oedema. Intradialytic hypotension is common affecting 30-40% of treatments and is consistently associated with at least a 30% increase in mortality and reduced quality-of-life. These dynamic changes in Blood Pressure (BP) and perfusion might be associated with altered cognition but the data are sparse and conflicting, possibly reflecting differences in study design; such as different methods and timings for cognitive assessments. Several small studies show cognitive function is best immediately before haemodialysis, worse during haemodialysis and improves the day after with a possible link to sudden fluid removal . Our own experience, using the Montreal Cognitive Assessment in 100 haemodialysis patients also showed cognitive decline during haemodialysis. A recent retrospective study of 121,000 patients report that peritoneal dialysis is associated with a 26% lesser-adjusted risk of newly diagnosed dementia compared to haemodialysis. One plausible mechanism of that benefit is that peritoneal dialysis does not cause sudden reductions in blood pressure.

Absence of intradialytic hypotension is emerging as a novel treatment goal 30. One possible way to prevent hypotension is to increase treatment time or frequency to allow more gentle fluid removal. A clinical trial of 245 patients showed 6 times weekly haemodialysis improved physical health scores whilst reducing intradialytic hypotension, fluid gains and left ventricular mass. A preliminary repeated measures study of 12 patients showed extended overnight haemodialysis was associated with improved cognitive function scores. These data are encouraging but come at the expense of increased treatment complications, cost and are currently unfeasible in most UK centres and worldwide. The use of cooler dialysate (34-35°C) to prevent intradialytic hypotension was first described in 1981. However, this therapy remains greatly underused because of perceptions about thermal symptoms. Cooler dialysate doesn't necessarily lower core-temperature and it is thought to prevent intradialytic hypotension by preventing a rise in core temperature and subsequent systemic vasodilation. A recent systematic review of cooler dialysate analyzed 26 trials in 484 patients. Compared with standard temperature dialysis, cooler dialysis reduced the rate of intradialytic hypotension by 70% (95% CI, 49-89%). Confidence in the estimates was limited by small sample sizes, attrition and a lack of appropriate blinding with no trial reporting long-term outcomes. A recent RfPB grant funded pilot clinical trial in 38 patients, showed lower temperature of dialysis fluid prevented the progression of ischemic brain white matter changes after one year which appeared to be linked to hemodynamic stability. The same trial also reported cooler dialysis fluid improved cardiac structure and function .

The effects of cooler dialysate on cognitive impairment, quality-of-life and illness burden have not been robustly tested or are not known. How well tolerated cooler dialysis fluid is also not well reported. A recent editorial called for larger trials using this cheap and universally applicable intervention that focused on these patient important outcomes. The current low usage of cooler dialysate in the UK affords an opportunity to definitively test this simple modification to haemodialysis as a potential intervention to prevent cognitive dysfunction and quality-of-life. There are several uncertainties around study design of a definitive trial of cooler dialysate and cognitive impairment, hence the need to formally assess these in a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged >18 years.
2. Receiving haemodialysis three (3) times per week for ESKD, for at least 3 months
3. Having proven mental capacity to understand the study and give informed consent

Exclusion Criteria:

1. Established diagnosis of dementia in a memory clinic or specialised service.
2. Receiving Acetylcholine Esterase Inhibitors
3. Receiving antipsychotic or antidepressants unless stable on treatment for at least 6 weeks
4. Current participation in a study of an investigational medicinal product
5. Inter-current infection
6. An operation date for a living donor kidney transplant within the period of the trial
7. Patients expected to survive less than 1 year according to the treating nephrologist
8. Patients prone to intra-dialytic hypotension or cardiovascular instability during haemodialysis according to the treating nephrologist
9. Patients who are currently taking triptans, dopamine antagonists, tramadol, sedative and opioid analgesics
10. Patients who have a known diagnosis or have other psychiatric conditions, including severe depression, bipolar affective disorder, severe anxiety, panic disorder, substance misuse or psychosis.
11. Currently involved in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Investigation of lower temperatures of dialysis and cognitive decline | 1.5 years
  To assess whether lower temperatures of dialysis fluid prevents the decline in cognitive function via utilisation of the Montreal Cognitive Assessment (MOCA) v7.2. The MOCA includes activities relating to Visuospatial / Executive (score out of 5); Naming (score out of 3); Memory (score of of 10); Attention (score out of 6); Naming (score out of 3) Abstraction (score out of 2); Delayed Recall (score out of 5) and Orientation (score out of 6). 1 point is given for each correct answer, and a higher score represents normal cognitive function, whilst lower scores represent possible cognitive decline. A total of 30 points can be achieved.

SECONDARY OUTCOMES:
Frequency of intradialytic hypotension | 1.5 years
  To measure the frequency of intradialytic hypotension as an explanatory outcome
Recruitment rates | 1.5 years
  To measure recruitment to inform the design of a larger clinical trial
Attrition Rates | 1.5 years
  To measure attrition rates to inform the design of a larger clinical trial
Non-recruitment reasons | 1.5 years
  To record reasons for non-recruitment and study attrition to inform the design of a larger clinical trial.
Depression rates | 1.5 years
  To measure depression in targeted population to be able to estimate exclusion rates of patients who would be suffering from "Depressive Pseudo Cognitive Impairment" from the future trial
Outcomes from Burden questionnaire to assess burden in patients and carers | 1.5 years
  To assess the burden of study-related interventions and assessments on patients and carers
Cognitive battery outcome | 1.5 years
  To assess the administration, suitability and adherence of the chosen cognitive method for patients, especially those from ethnic minorities
Carers Burden assessment | 1.5 years
  To assess the administration and suitability of the chosen method for measuring carers' burden in this group.
Quality Of Life outcomes | 1.5 years
  To assess the administration and suitability of the Assessment of Quality of Life 6 (AQoL-6) for quality of life measures and activities of daily living in haemodialysis participants. The AQoL-6 is a likert scale ranging from 'Never' (=1), 'Rarely' (=2) 'Some of the Time' (=3) 'Often' (=4) and 'Nearly All of the Time' (=5) - there are 20 items so a total score of 100 can be obtained. A score of 100 represents very poor quality of life, where as a score of 0 indicates very good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: George Tadros, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasgupta I, Odudu A, Baharani J, Fergusson N, Griffiths H, Harrison J, Hameed A, Maruff P, Ryan L, Thomas N, Woodhall G, Tadros G. Evaluation of effect of cooled haemodialysis on cognition in patients with end-stage kidney disease (ECHECKED) feasibility randomised controlled trial results. BMC Nephrol. 2024 Dec 19;25(1):466. doi: 10.1186/s12882-024-03883-6. PMID 39702060
- [Derived] Kulkarni M, Prabhu AR, Rao IR, Nagaraju SP. Interventions for preventing haemodialysis dysequilibrium syndrome. Cochrane Database Syst Rev. 2024 May 22;5(5):CD015526. doi: 10.1002/14651858.CD015526.pub2. PMID 38775299
- [Derived] Dasgupta I, Odudu A, Baharani J, Fergusson N, Griffiths H, Harrison J, Maruff P, Thomas GN, Woodhall G, Youseff S, Tadros G. Evaluation of the effect of Cooled HaEmodialysis on Cognitive function in patients suffering with end-stage KidnEy Disease (E-CHECKED): feasibility randomised control trial protocol. Trials. 2020 Sep 30;21(1):820. doi: 10.1186/s13063-020-04725-0. PMID 32998761